CLINICAL TRIAL: NCT04276545
Title: Dexmedetomidine Improves the Surgical Field and Postoperative Recovery of Nasal Endoscopic Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Jinhong Wu, Attending anesthesiologist, Eye & ENT Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: EyeEntFudan2
Record Dates: First submitted 2020-02-09; First posted 2020-02-19 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Dexmedetomidine; Bleeding; Surgical Field
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IV administration of dexmedetomidine (Experimental): IV administration of a single loading dose DEX (0.5μg/kg)
  Interventions: Drug: IV administration of DEX to investigate the effects for functional nasal endoscopic surgery; Drug: IV administration of Midazolam to investigate the effects for functional nasal endoscopic surgery
- IV administration of midazolam (Active Comparator): IV administration of midazolam (0.05mg/kg)
  Interventions: Drug: IV administration of DEX to investigate the effects for functional nasal endoscopic surgery; Drug: IV administration of Midazolam to investigate the effects for functional nasal endoscopic surgery

INTERVENTIONS:
Drug: IV administration of DEX to investigate the effects for functional nasal endoscopic surgery — IV administration of a single loading dose DEX (0.5μg/kg) after induction within 10 minutes.
Drug: IV administration of Midazolam to investigate the effects for functional nasal endoscopic surgery — IV administration of midazolam (0.05mg/kg) after induction.

SUMMARY:
Studies showed dexmedetomidine (DEX) could improve surgical field, but the effect for functional nasal endoscopic surgery (FESS) was unclear. The investigators explored IV administration of a single loading dose DEX (0.5μg/kg) for FESS, and IV administration of midazolam (0.05mg/kg) as a control with comparision of surgical field, haemodynamics, ventilation parameters and recovery.

DETAILED DESCRIPTION:
The participants received an induction of anesthesia with propofol 2-3 mg/kg, sufentanyl 0.2 μg/kg, and rocuronium 0.6 mg/kg, and then insertion of a flexible laryngeal mask airway was conducted using the index finger insertion technique by anesthesia providers with a minimum of four years endotracheal intubation experience. Mechanical ventilation parameters were as follows: pressure-controlled ventilation mode, ventilation pressure: 12, respiratory rate: 12, oxygen concentration: 50%. The maintenance of general anesthesia was performed with sevoflurane at minimum alveolar concentration of 1.3. After induction, a single loading dose DEX (0.5μg/kg) was IV infusion within 10 minutes, or IV administration of midazolam (0.05mg/kg). Heart rate, blood pressure, tidal volume, ventilation pressure and ETCO2 after insertion of a LMA, 10 minutes, 20 minutes, 30 minutes after drug infusion and transferred to PACU, besides heart rate and blood pressure were recorded before and after induction. Surgical field was evaluated at the time of 10 minutes and 20 minutes after drug infusion. Blood gas analysis was performed just transferred to PACU and before transferred to ward.

ELIGIBILITY:
Inclusion Criteria:

* 120 participants who diagnosed with nasosinusitis
* The participants need undergo functional nasal endoscopic surgery
* The participants signed the informed consent

Exclusion Criteria:

* The participants were excluded with any diseases about respiration, circulation, liver and kidney
* The participants were rejected of the consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of surgical field according to the scale reported by Boezaart A.P. in the two groups | Through study completion, an average of 1 year
  Levels of the scale reported by Boezaart A.P. as follows:
  0. No bleeding.
  1. Slight bleeding - no suctioning of blood required.
  2. Slight bleeding - occasional suctioning required. Surgical field not threatened.
  3. Slight bleeding - frequent suctioning required. Bleeding threatens surgical field a few seconds after suction is removed.
  4. Moderate bleeding - frequent suctioning required. Bleeding threatens surgical field directly after suction is removed.
  5. Severe bleeding - constant suctioning required. Bleeding appears faster than can be removed by suction. Surgical field severely threatened and surgery not possible.
  Evaluation of surgical field was carried out by Kruskal-Wallis H test.

SECONDARY OUTCOMES:
Comparision of heart rate and mean blood pressure during anesthesia in the two groups | Through study completion, an average of 1 year
  Heart rate (beats/minutes) and mean blood pressure (mmHg) were recorded every 10 minutes, and analyzed with Student's t-test
Comparision of recovery time and blood gas analysis in PACU in the two groups | Through study completion, an average of 1 year
  Recovery time (minutes) included from entering to leaving PACU, and blood gas analysis just before leaving PACU

CONTACTS AND LOCATIONS:
Overall Officials: Shenghai Zhang, Study Director — Eye, Ear, Nose and Throat Hospital, Fudan University
Locations (1):
- Eye, Ear, Nose and Throat Hospital, Shanghai, Shanghai Municipality, China